CLINICAL TRIAL: NCT05212532
Title: A Proof-of-Concept Study Evaluating Safety, Tolerability, and Preliminary Efficacy of EOM613 in COVID-19 Infected Patients With Severe Symptoms
Brief Title: A Proof-of-Concept Study Evaluating EOM613 in COVID-19 Infected Patients With Severe Symptoms
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: EOM Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL-EOM613-001
Record Dates: First submitted 2021-08-25; First posted 2022-01-28 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: COVID-19 Pneumonia; COVID-19 Respiratory Infection; COVID-19 Acute Respiratory Distress Syndrome
Keywords: Cytokines; Chemokines; COVID-19; SARS-CoV-2; Immune modulation
MeSH Terms: conditions — COVID-19 | interventions — EOM613

STUDY DESIGN:
Intervention Model Description: Open label study will include 2 cohorts, non-ICU hospitalized and ICU hospitalized patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non-ICU hospitalized (Experimental): Patients who are hospitalized at study enrollment but are not being treated in the ICU
  Interventions: Drug: EOM613
- ICU hospitalized (Experimental): Patients who, at study enrollment, are being treated in the hospital ICU
  Interventions: Drug: EOM613

INTERVENTIONS:
Drug: EOM613 — peptide nucleic acid (PNA)

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and preliminary efficacy of EOM613, a peptide nucleic acid with novel immune-modulating properties, in treating patients with severe COVID-19 infections. This proof-of-concept study is the first clinical trial of EOM613 in this patient population.

DETAILED DESCRIPTION:
Much of the morbidity and mortality in COVID-19 infection is thought to be the result of an overly zealous attack by the immune system (e.g., cytokine storm and IL-6 elevations) as it attempts to counteract the viral infection. Some drugs with immunomodulatory effects (e.g., dexamethasone, tocilizumab) have been shown to reduce virus-induced cytokine storms and key pro-inflammatory cytokines, including IL-6.

EOM613 is a peptide nucleic acid with novel immune-modulating properties, including modulation of IL-6 expression. It has an excellent safety profile and has yielded promising therapeutic results in patients with Acquired Immunodeficiency Syndrome (AIDS), cancer cachexia and severe rheumatoid arthritis. EOM613 was reported to have antiviral activity in cell cultures inoculated with Human Immunodeficiency Virus (HIV) or adenovirus. This proof-of-concept study is the first clinical trial of EOM613 in patients with COVID-19 infection.

This study will include two cohorts of hospitalized patients, non-ICU and ICU. In non-ICU patients, EOM613 is to be administered subcutaneously (SC) at a dose of 2 mL once daily (QD) for 10 days, for a total of 20 mL. In ICU patients, EOM613 is to be administered SC at a dose of 2 mL twice daily (BID) for 5 days followed by 2 mL QD for 5 days, for a total of 30 mL.

The primary objective and outcome measures include assessment of safety and tolerability of EOM613, based on clinical laboratory, physical exams, and assessment of adverse events (AEs). The secondary objectives and outcome measures are 1) The proportions of non-ICU patients discharged with and without progression to invasive mechanical ventilation or ICU; 2) The proportion of ICU patients who die, are discharged to the infirmary, or discharged from the hospital; and 3) Assessment of levels of pro- and anti-inflammatory cytokines in Cytokine Panel 13, and their correlations with primary and secondary endpoints.

ELIGIBILITY:
1. Inclusion Criteria

   1. Non-ICU cohort:

      * Males or females ≥18 years and < 85 years of age
      * Positive test for Severe Acute Respiratory Syndrome Coronavirus 2 (SARS- CoV-2) by nasopharyngeal sampling using a reliable nucleic acid Reverse Transcription-Polymerase Chain Reaction (RT-PCR) assay or fast serological tests confirmed by RT PCR afterward
      * Hospitalized for Acute Respiratory Distress Syndrome (ARDS) or pneumonia
      * Requires oxygen therapy by nasal catheter or mask, but not invasive mechanical ventilation at the enrollment
   2. ICU cohort:

      * Males or females ≥18 years and < 85 years of age
      * Positive test for SARS-CoV-2 by nasopharyngeal sampling using a reliable nucleic acid RT-PCR assay
      * Hospitalized for ARDS or pneumonia and requires invasive mechanical ventilation at enrollment
   3. Both cohorts:

      * Participant or suitable proxy able to provide written informed consent before study procedures are performed
      * Able to adhere to the study schedule and other protocol requirements
      * No known contraindications for administering EOM613, including Mycobacterium tuberculosis infection (assessed by the anamnesis) or receiving immunosuppressant therapy after transplant
      * Not enrolled in another study of an investigational agent during this study
      * Patients who developed complications of COVID-19 (such as myocardial disease, kidney dysfunction, clotting disorder, encephalitis, severe fatigue, or multi-immune inflammatory syndrome) are eligible
2. Exclusion Criteria

   1. Both cohorts:

      * Active participation in any other clinical trial of an experimental treatment for COVID-19
      * Participation in another clinical trial with any investigational new drug within 12 months before enrollment, except if there is a possible benefit to the participant in the investigator's opinion (According to the Brazilian Resolution CNS 251/97 II.2-J)
      * Concurrent treatment with other agents with actual or possible direct-acting antiviral activity against SARS-CoV-2 is prohibited <24 hours before study medication initiation
      * Sequential Organ Failure Assessment Score >10
      * Stage 4 severe chronic kidney disease or requiring dialysis (i.e., estimated Glomerular Filtration Rate [eGFR] <30)
      * Active cancer receiving any therapeutic intervention or under palliative care
   2. Both cohorts, conditions existing before COVID-19:

      * Chronic Obstructive Pulmonary Disease (COPD)
      * Heart failure or cardiomyopathies
      * Sickle cell disease
      * Solid-organ transplantation
      * Uncontrolled or poorly controlled Type 2 diabetes mellitus
      * Immunodeficiency or immunosuppressive therapy
      * Pregnant or breastfeeding
      * Consideration by the investigator, for any reason, that the subject is an unsuitable candidate to receive study treatment
      * Known active Mycobacterium tuberculosis infection (assessed by the anamnesis)
      * Patients who are unwilling or unable to follow protocol requirements
      * Patients with body mass index (BMI) < 18 kg/m2 or > 40 kg/m2

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-08-09 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to day 11 in mean blood urea nitrogen (BUN) level. | Baseline and day 11 or discharge, whichever comes first.
  The BUN primary outcome measure is its change from baseline to day 11 or to discharge, whichever comes first (BUN is also assessed on days 2, 5, and 8). BUN is obtained from a venous blood draw and measured in millimoles of urea per liter. 2.1 to 8.5 mmol/L is considered normal; values above 8.5 mmol/L may indicate renal impairment.
Change from baseline to day 11 in mean blood creatinine level. | Baseline and day 11 or discharge, whichever comes first.
  The blood creatinine primary outcome measure is its change from baseline to day 11 or to discharge, whichever comes first (blood creatinine is also assessed on days 2, 5, and 8). Blood creatinine is obtained from a venous blood draw and measured in micromoles of creatinine per liter. 65.4 to 119.3 micromoles/L in adult women and 52.2 to 91.9 micromoles/L in adult men are considered normal; values above these ranges may indicate renal impairment.
Change from baseline to day 11 in mean blood lymphocyte count. | Baseline and day 11 or discharge, whichever comes first.
  The blood lymphocyte count primary outcome measure is its change from baseline to day 11 or to discharge, whichever comes first (blood lymphocyte count is also assessed on days 2, 5, and 8). Blood lymphocyte count is obtained from a venous blood draw and measured as the number of lymphocytes per microliter of blood. Between 1,000 and 3000 lymphocytes per microliter of blood is considered normal. Values below this range have correlated with the severity of COVID-19 infection; values above this range can be indicative of an infection, cancer of the blood or lymphatic system, or an autoimmune disorder.
Change from baseline to day 11 in mean serum soluble interleukin-2 receptor (sIL-2R) level. | Baseline and day 11 or discharge, whichever comes first.
  The serum sIL-2R primary outcome measure is its change from baseline to day 11 or to discharge, whichever comes first (serum sIL-2R will also be assessed on days 2, 5, 8, 14 and 28). Serum sIL-2R levels are measured with a Quantitative Multiplex Bead Assay. The normal range has been reported as 175.3 - 858.2 pg/mL. Elevated levels are found in individuals with severe inflammatory conditions and solid tumors.
Change from baseline to day 11 in mean serum interleukin-6 (IL-6). | Baseline and day 11 or discharge, whichever comes first.
  The serum IL-6 primary outcome measure is its change from baseline to day 11 or to discharge, whichever comes first (serum IL-6 will also be assessed on days 2, 5, 8, 14 and 28). Serum IL-6 levels are measured with a Quantitative Multiplex Bead Assay. Normal values have been reported as <2.0 pg/mL. Elevated levels are associated with inflammatory conditions and predict lower chances of survival in COVID-19 patients.
Change from baseline to day 11 in mean serum interleukin-10 (IL-10) levels. | Baseline and day 11 or discharge, whichever comes first.
  The serum IL-10 primary outcome measure is its change from baseline to day 11 or discharge, whichever comes first (serum IL-10 will also be assessed on days 2, 5, 8, 14 and 28). Serum IL-10 levels are measured with a Quantitative Multiplex Bead Assay. Normal values have been reported as <2.8 pg/mL. Elevated levels are associated with inflammatory conditions and predict lower chances of survival in COVID-19 patients.

SECONDARY OUTCOMES:
Median change from baseline to day 56 in World Health Organization (WHO) Scale Assessment of COVID-19 Symptom Severity | Baseline and day 56 or death, whichever comes first
  The WHO Scale secondary outcome measure is the median change from baseline to day 56. This ordinal Scale is from 0 (no clinical/virological evidence of infection) to 8 (death). Scale assessments are made on patients on days 1-14, 21, 28, 42 and 56. Scale assessments of discharged patients are made during a home visit by a study nurse.
Percent of hospital days with ventilator and/or oxygen use, and percent of hospital days with maximum ventilator pressure and maximum oxygen use | Day 1 (baseline) of ventilator and/or oxygen use until ventilator and/or oxygen use is discontinued
  Daily recording of ventilator and oxygen use (on or off), ventilator pressure, and oxygen use (percent and flow rate) in the morning and evening for patients requiring respiratory assistance. These data will be used to calculate the mean percent of total hospital days with ventilator and/or oxygen use, and the mean percent of days of maximum ventilator pressure and maximum oxygen use from day 1 of ventilator and/or oxygen use to subsequent days.

CONTACTS AND LOCATIONS:
Overall Officials: Irach Taraporewala, PhD, Study Chair — CEO and Director, EOM Pharma; Frank L Douglas, PhD, MD, Study Director — Scientific Advisor & Chair of Scientific Advisory Board, EOM Pharma; Florentino Cardoso Filho, MD, PhD, Principal Investigator — Physician, Casa de Saude Hospital, Campinas, SP
Locations (4):
- Brazil (4):
  - Oswaldo Cruz, Manguinhos, Rio de Janeiro
  - Hospital de Amor, Barretos, São Paulo
  - Hospital Municipal de Barueri, Barueri, São Paulo
  - Casa De Saúde, Boqueirão, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Advanced Viral Research Corp. (ADVR). ADVR reports AVR118 inhibits inflammatory arthritis in animal model and in rheumatoid arthritis patients in human clinical trial. ADVR press release, PR Newswire, December 3, 2003.
- [Background] Chasen M, Bhargava R, Hirschman SZ, Taraporewala I. Phase II study of OHR/AVR118 in anorexia- cachexia. Abstract of poster presentation at the 7th Cachexia conference, Kobe/Osaka, Japan, December 9-11, 2013. J Cachexia Sarcopenia Muscle 2013;4(4):335-6.
- [Background] Chasen M, Hirschman SZ, Bhargava R. Phase II study of the novel peptide-nucleic acid OHR118 in the management of cancer-related anorexia/cachexia. J Am Med Dir Assoc. 2011 Jan;12(1):62-7. doi: 10.1016/j.jamda.2010.02.012. Epub 2010 May 15. PMID 21194662
- [Background] COVID-19 Treatment Guidelines, Interleukin-6 Inhibitors. National Institutes of Health. https://www.covid19treatmentguidelines.nih.gov/therapies/immunomodulators/interleukin-6-inhibitors/. Updated April 21, 2021. Accessed August 24, 2021.
- [Background] Diao L, Meibohm B. Pharmacokinetics and pharmacokinetic-pharmacodynamic correlations of therapeutic peptides. Clin Pharmacokinet. 2013 Oct;52(10):855-68. doi: 10.1007/s40262-013-0079-0. PMID 23719681
- [Background] D'Olimpio JT, Chasen MR, Sharma R, Diego M, Gullo V, MacDonald N. Phase II study of AVR118 in the management of cancer-related anorexia/cachexia. Doi: 10.1200/jco.2009.27.15_suppl.e20631 (abstract presentation). Journal of Clinical Oncology 2009; 27, No. 15_suppl., e20631-e20631.
- [Background] D'Olimpio JT, Hirschman SZ, Shtemer Z, Didiego M. Anti-cachectic effects of a novel peptide nucleic acid: Preliminary results of a phase I/II clinical trial. Doi: 10.1200/jco.2004.22.90140.8087 (abstract presentation). Journal of Clinical Oncology. July 15, 2004; 22, no. 14_suppl 8087-8087.
- [Background] Friedland B. In vitro antiviral activity of a peptide-nucleic acid solution against the human immunodeficiency virus and influenza A virus. J R Soc Health. 1991 Oct;111(5):170-1. doi: 10.1177/146642409111100505. PMID 1724467
- [Background] Hirschman SZ, Chen CW. Peptide nucleic acids stimulate gamma interferon and inhibit the replication of the human immunodeficiency virus. J Investig Med. 1996 Aug;44(6):347-51. PMID 8795297
- [Background] Hirschman SZ. Activation of human monocytes/macrophages by OHR/AVR118 promotes both pro-and anti-inflammatory phenotypes. Available: https://www.scirp.org/journal/PaperInformation.aspx?paperID=42617. Accessed August 24, 2021. Adv Bioscience Biotechnology. 2014, 5:161-168.
- [Background] Hojyo S, Uchida M, Tanaka K, Hasebe R, Tanaka Y, Murakami M, Hirano T. How COVID-19 induces cytokine storm with high mortality. Inflamm Regen. 2020 Oct 1;40:37. doi: 10.1186/s41232-020-00146-3. eCollection 2020. PMID 33014208
- [Background] Lazzarino DA, Diego M, Musi E, Hirschman SZ, Alexander RJ. CXCR4 and CCR5 expression by H9 T-cells is downregulated by a peptide-nucleic acid immunomodulator. Immunol Lett. 2000 Nov 1;74(3):189-95. doi: 10.1016/s0165-2478(00)00258-3. PMID 11064099
- [Background] Lazzarino DA, de Diego M, Hirschman SZ, Zhang KY, Shaikh S, Musi E, Liaw L, Alexander RJ. IL-8 and MCP-1 secretion is enhanced by the peptide-nucleic acid immunomodulator, Product R, in U937 cells and primary human monocytes. Cytokine. 2001 May 21;14(4):234-9. doi: 10.1006/cyto.2001.0867. PMID 11448124
- [Background] Levett PN, Hirschman SZ, Roach TC, Broome H, Alexander RJ, Fraser HS. Randomized, placebo-controlled trial of product R, a peptide-nucleic acid immunomodulator, in the treatment of adults infected with HIV. HIV Clin Trials. 2002 Jul-Aug;3(4):272-8. doi: 10.1310/N34A-653T-ABF5-8Q1R. PMID 12187500
- [Background] Scherger S, Henao-Martinez A, Franco-Paredes C, Shapiro L. Rethinking interleukin-6 blockade for treatment of COVID-19. Med Hypotheses. 2020 Nov;144:110053. doi: 10.1016/j.mehy.2020.110053. Epub 2020 Jun 27. PMID 32758889
- [Background] Alexander R.J., Meyer K.A., Camposano E., Lazzarino D.A., De Diego M. Product R induces differentiation of the human myelocytic leukemia cell line HL-60. American Association for Cancer Research Special Conference (Proteases, Extracellular Matrix and Cancer). Hilton Head Island, SC, USA, 2002.